CLINICAL TRIAL: NCT05435586
Title: The Effect of Digital Game Supported Web Based Breastfeeding Education and Counseling on Breastfeeding Self-Efficacy, Breastfeeding Success and Breast Problems: A Randomized Controlled Study
Brief Title: Digital Game Supported Breastfeeding Self-Efficacy, Breastfeeding Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Özlem Ülkü BULUT, Lecturer, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Oyunlastirmailemzirme
Record Dates: First submitted 2022-06-01; First posted 2022-06-28 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Self Efficacy; Breast Feeding, Exclusive
Keywords: gamification; breastfeeding self-efficacy; breastfeeding success; breast problems
MeSH Terms: conditions — Breast Feeding | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: The study is an experimental study with pretest-posttest parallel group randomized controlled.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The research data were collected on a web-based platform by the researcher, who did not know who was in the experimental and control groups, and transferred to the computer by someone else. A statistician analyzed the coded data in groups. Statistical analyzes have been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web Based Breastfeeding Education and Counseling with Digital Game Support (Experimental): During pregnancy;
  * Application of the "Individual and Obstetrical Characteristics Evaluation Form of Pregnant Women" and "Breastfeeding Self-Efficacy Scale Antenatal Form" (Pre-Test).(32-34 weeks of gestation)
  * Program will be applied to 30 women at 35-37 gestational weeks.
  * Breastfeeding Self-Efficacy Scale (Antenatal form) will be applied to at the end of 37th gestational week.
  In the postpartum period;
  * The LATCH Breastfeeding Diagnostic Tool and Breastfeeding Assessment Scale (IBFAT) will be administered on the first postpartum day.
  * Program will be applied to 30 women during the first 2 weeks postpartum.
  * At the end of the postpartum 2nd week, Breastfeeding Behavior and Breast Problems Evaluation Form will be administered.
  * Breastfeeding Self-Efficacy Scale (Postpartum form) and Breast Problems Evaluation form will be administered at postpartum 8th week.
  Interventions: Other: Web Based Breastfeeding Education and Counseling with Digital Game Support
- Standardized breastfeeding education (No Intervention): During pregnancy;
  * Application of the "Individual and Obstetrical Characteristics Evaluation Form of Pregnant Women" and "Breastfeeding Self-Efficacy Scale Antenatal Form" (Pre-Test).(32-34 weeks of gestation)
  * 30 women will receive the routine care applied during pregnancy in the hospital.
  * At the end of the 37th week, the Breastfeeding Self-Efficacy Scale (Antenatal form) will be administered to the women in the control group.
  In the postpartum period;
  * 30 women will receive the standard breastfeeding training in the hospital.
  * The LATCH Breastfeeding Diagnostic Tool and Breastfeeding Assessment Scale (IBFAT) will be administered on the first postpartum day.
  * At the end of the postpartum 2nd week, the Breastfeeding Behavior and Breast Problems Evaluation Form will be applied.
  * Breastfeeding Self-Efficacy Scale (Postpartum form) and Breastfeeding Behavior and Breast Problems Evaluation Form will be administered at the postpartum 8th week.

INTERVENTIONS:
Other: Web Based Breastfeeding Education and Counseling with Digital Game Support — The educational content prepared by the researcher on the web page will be integrated into the game program designed with the gamification technique. In this designed program, users will be notified at appropriate times to enter the system and play games from the link sent via e-mail. After the users have finished the game, they will fill the scale in the relevant week and will only be able to exit the system in that way.
  Other Names: Gamification
  Arms: Web Based Breastfeeding Education and Counseling with Digital Game Support

SUMMARY:
Purpose: This study will be conducted to determine the effect of digital game supported web-based breastfeeding education and counseling on breastfeeding self-efficacy, breastfeeding success and breast problems.

Method: This is an experimental study with a randomized controlled pretest-posttest parallel group, and 30 women will be included in the experimental group and 30 women in the control group. In the study, Pregnant Women's Individual and Obstetric Characteristics Evaluation Form, Breastfeeding Self-Efficacy Scale Short Form (EÖYÖ), LATCH Breastfeeding Assessment Tool, Breastfeeding Evaluation Scale (IBFAT), Breastfeeding Behavior and Breast Problems Evaluation Form will be used. The data will be analyzed in SPSS program.

In the Digital Game Supported Web-Based Breastfeeding Education and Counseling Program, the educational content prepared by the researcher will be integrated into the game program designed with the gamification technique. An education program will be applied to the women in the experimental group during pregnancy and postpartum period. Women in the control group will receive the standard breastfeeding training in the hospital. Measurement tools will be applied to all participants for a total of three times, once before birth and twice after birth.

Conclusion and Suggestions: In this planned study, it was aimed to teach women about breastfeeding in a digital environment in a fun way. It is thought that web-based breastfeeding education and counseling supported by digital games will have a positive effect on breastfeeding self-efficacy, breastfeeding success and breast problems.

DETAILED DESCRIPTION:
Breastfeeding has an important place in the healthy development of the baby, maternal benefits and mother-infant bonding. One of the most important factors affecting breastfeeding duration and success is the mother's perception of breastfeeding self-efficacy. In order to increase breastfeeding success and self-efficacy, it is very important for women to know about breastfeeding and the problems they may encounter. In the digital age, online training or access to online materials is easy and effortless. In the learning method with gamification, which has an important place in digital education, the behavior style that is intended to be taught to individuals can be taught more effectively and easily in accordance with the learning objectives. The inclusion and use of gamified features in web-based health interventions is known to increase user experience, increasing interest and fun.

In this study, it is thought that the Digital Game Supported Web-Based Breastfeeding Education and Counseling Program, which will be applied as individual sessions to women starting from the prenatal period until the postpartum 2nd month, will have positive effects on breastfeeding self-efficacy, breastfeeding success and breast problems. It is estimated that these results can guide professionals working with mothers and babies in the field and make a unique contribution to the field.

ELIGIBILITY:
Inclusion Criteria:

* Primipara,
* 32-36. between gestational weeks,
* Those who have not received a planned breastfeeding training before,
* Speaking and understanding Turkish,
* Women with a smart phone/tablet/computer with internet connection will be included in the study.

Exclusion Criteria:

* Having a chronic disease,
* Those who will give birth by planned cesarean section,
* Breastfeeding contraindications
* Women with risky pregnancies will not be included in the study.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale Short Form Antenatal score | "pre-intervention"
  Breastfeeding Self-Efficacy Scale was developed by Dennis in 1999 and consists of 33 items. Later, the scale was reduced to 14 items by Dennis in 2003 and the Breastfeeding Self-Efficacy Scale Short Form was developed. The Turkish validity and reliability of the Breastfeeding Self-Efficacy Scale Short form was performed by Aluş Tokat and Okumus in 2009. This scale assesses how competent mothers feel about breastfeeding. The scale consists of 14 items and includes a 5-point Likert-type evaluation consisting of Not sure at all: 1, Not very sure: 2, Sometimes I am sure: 3, I am sure: 4, Very sure: 5 options. The lowest score that can be obtained from the entire scale is 14 and the highest score is 70. A high score from the scale indicates a high perception of breastfeeding self-efficacy.
Breastfeeding Self-Efficacy Scale Short Form Antenatal score | "At the end of 37th gestational week."
  Breastfeeding Self-Efficacy Scale was developed by Dennis in 1999 and consists of 33 items. Later, the scale was reduced to 14 items by Dennis in 2003 and the Breastfeeding Self-Efficacy Scale Short Form was developed. The Turkish validity and reliability of the Breastfeeding Self-Efficacy Scale Short form was performed by Aluş Tokat and Okumus in 2009. This scale assesses how competent mothers feel about breastfeeding. The scale consists of 14 items and includes a 5-point Likert-type evaluation consisting of Not sure at all: 1, Not very sure: 2, Sometimes I am sure: 3, I am sure: 4, Very sure: 5 options. The lowest score that can be obtained from the entire scale is 14 and the highest score is 70. A high score from the scale indicates a high perception of breastfeeding self-efficacy.
The Infant Breastfeeding Assesment Tool score | "First day postpartum"
  The Infant Breastfeeding Assesment Tool (IBFAT) It was developed by Mary Kay Matthews in 1988. The scale is a measurement tool developed to determine temporary feeding difficulties in the first 4 to 5 days in healthy and term babies. The Turkish validity and reliability study of the scale was carried out by Çelik and Demirci, and the Cronbach alpha coefficient was calculated as 0.92 in this study. The scale consists of six questions and the evaluation is made by the mothers. Scoring is done on the basis of the mothers' answers to the questions.
  The first question in the scale is about the baby's feeding status (deep sleep, sleepy, calm awake, crying). In the last question, mothers are asked to state their feelings during feeding (Very satisfied, satisfied, not very satisfied, not satisfied). These two questions are not included in the scoring and are evaluated separately.
The LATCH Breastfeeding Diagnostic Tool | "First day postpartum"
  The LATCH Breastfeeding Diagnostic Tool It was developed by Mary Kay Matthews in 1988. The scale is a measurement tool developed to determine temporary feeding difficulties in the first 4 to 5 days in healthy and term babies. The Turkish validity and reliability study of the scale was carried out by Çelik and Demirci, and the Cronbach alpha coefficient was calculated as 0.92 in this study. The scale consists of six questions and the evaluation is made by the mothers. Scoring is done on the basis of the mothers' answers to the questions.
  The first question in the scale is about the baby's feeding status (deep sleep, sleepy, calm awake, crying). In the last question, mothers are asked to state their feelings during feeding (Very satisfied, satisfied, not very satisfied, not satisfied). These two questions are not included in the scoring and are evaluated separately.
Breastfeeding Self-Efficacy Scale Short Form Postnatal score | "8 weeks postpartum"
  Breastfeeding Self-Efficacy Scale was developed by Dennis in 1999 and consists of 33 items. Later, the scale was reduced to 14 items by Dennis in 2003 and the Breastfeeding Self-Efficacy Scale Short Form was developed. The Turkish validity and reliability of the Breastfeeding Self-Efficacy Scale Short form was performed by Aluş Tokat and Okumus in 2009. This scale assesses how competent mothers feel about breastfeeding. The scale consists of 14 items and includes a 5-point Likert-type evaluation consisting of Not sure at all: 1, Not very sure: 2, Sometimes I am sure: 3, I am sure: 4, Very sure: 5 options. The lowest score that can be obtained from the entire scale is 14 and the highest score is 70. A high score from the scale indicates a high perception of breastfeeding self-efficacy.

SECONDARY OUTCOMES:
Breastfeeding Behavior and Breast Problems Evaluation Form | "2 weeks postpartum"
  The Breastfeeding Behavior and Breast Problems Evaluation Form, prepared by the researcher after a literature review, will be applied to the women in order to determine the breastfeeding behavior and breast problems of women in the postpartum period.
Breastfeeding Behavior and Breast Problems Evaluation Form | "8 weeks postpartum"
  The Breastfeeding Behavior and Breast Problems Evaluation Form, prepared by the researcher after a literature review, will be applied to the women in order to determine the breastfeeding behavior and breast problems of women in the postpartum period.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University Etlik Hospital, Ankara, Turkey (Türkiye)